CLINICAL TRIAL: NCT05634564
Title: Efficacy and Safety of Concurrent Chemoradiotherapy Combined With Immunotherapy in Patients With Potentially Resectable Pancreatic Cancer
Brief Title: Concurrent Chemoradiotherapy Combined With Immunotherapy in Patients With Potentially Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Du Juan, Clinical Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP-PC
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tislelizumab; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent radiochemotherapy combined with immunotherapy (Experimental): Participants will receive tislelizumab plus gemcitabine and nab-paclitaxel in cycles of 21 days. Non-progressors will plus concurrent radiotherapy during the 3rd cycle of chemotherapy. After 4-6 cycles treatment, Multiple disciplinary team (MDT) will evaluate whether to undergo radical surgery.
  Interventions: Drug: Tislelizumab; Drug: Gemcitabine; Drug: Nab paclitaxel; Radiation: Hypofractionated radiotherapy with simultaneous integrated boost

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg administered intravenously on Days 1 of every 3 weeks.
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 administered intravenously on Days 1 & 8 of every 3 weeks.
Drug: Nab paclitaxel — Gemcitabine 125 mg/m^2 administered intravenously on Days 1 & 8 of every 3 weeks.
Radiation: Hypofractionated radiotherapy with simultaneous integrated boost — Radiotherapy plan: Planning gross tumor volume (PGTV) 5Gy*10 fractions, Planning target volume (PTV) 3Gy*10 fractions.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy combined with immunotherapy in patients with potentially resectable pancreatic cancer.

DETAILED DESCRIPTION:
Due to the hidden onset and rapid progression of pancreatic cancer, most patients are already locally advanced or have distant metastasis at the time of diagnosis and lose the opportunity for surgery. Even among operable patients, about 50% will have recurrence and metastasis one year after surgery. Therefore, more and more evidence supports neoadjuvant therapy for patients with high risk factors for resectable pancreatic cancer, and conversion therapy followed by surgery for patients with borderline resectable and locally advanced pancreatic cancer. Therefore, the objective of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy combined with immunotherapy in patients with potentially resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years； 2. Eastern Cooperative Oncology Group (ECOG) score of 0-1; 2. Pancreatic cancer confirmed by histology or cytology; 3. Potentially resectable pancreatic cancer documented by contrast enhanced CT (or MRI) scan; 4. Hematological indexes: Neutrophil count >= 1.5 x 10^9/L Hemoglobin >= 10g / dl Platelet count >= 100 x 10^9 / L 5. Biochemical indicators: Total bilirubin <= 1.5 x upper limit of normal value (ULN); Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 1.5 x ULN; Creatinine clearance rate >= 60ml / min.

6. Participants of childbearing age need to take appropriate protective measures (contraceptive measures or other methods of birth control) before entering the group and during the test: 7. Signed informed consent; 8. Follow the protocol and follow-up procedures.

Exclusion Criteria:

1. Have received systematic anti-tumor treatment.
2. Previous history of other tumors, except for cervical cancer in situ, treated squamous cell carcinoma or bladder epithelial tumor (TA and TIS) or other malignant tumors that have received radical treatment (at least 5 years before enrollment).
3. Active bacterial or fungal infection (> = level 2 of National Cancer Institute Common Toxicity Criteria (NCI-CTC), Version 3.0).
4. Human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) infection, uncontrollable coronary artery disease or asthma, uncontrollable cerebrovascular disease or other diseases considered by researchers to be out of the group.
5. Autoimmune diseases or immune defects who are treated with immunosuppressive drugs.
6. Pregnant and lactating women. Pregnant women of childbearing age must be tested negative within 7 days before entering the group.
7. Drug abuse, clinical or psychological or social factors make informed consent or research implementation affected.
8. Allergic to programmed cell death protein-1 (PD-1) monoclonal antibody immunotherapy drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  RECIST Version 1.1

SECONDARY OUTCOMES:
R0 resection rate | Up to 1 years
  R0 resection rate
Median Progression Free Survival (mPFS) | Up to 2 years
  RECIST Version 1.1
Median Overall survival (mOS) | Up to 2 years
  RECIST Version 1.1
Disease control rate (DCR) | Up to 2 years
  RECIST Version 1.1
Pathological grade of tumor tissue after neoadjuvant therapy | Up to 1 years
  Pathological grade of tumor tissue after neoadjuvant therapy
Adverse Events | Up to 2 years
  Adverse event (AE)、Serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ni J, Sun Y, Cheng H, Bai X, Tong F, Zhang X, Wang X, Mao L, Li G, Shen S, Kong W, He J, Li A, Chen J, Tang M, Chen B, Li Q, Gu Q, Lu Z, Chen D, Sha H, Liu B, Qiu Y, Du J. Tislelizumab and hypofractionated radiotherapy plus nab-paclitaxel/gemcitabine as conversion therapy for BRPC/LAPC: A Phase II trial with dynamic biomarker monitoring. Clin Cancer Res. 2025 Dec 1. doi: 10.1158/1078-0432.CCR-25-2461. Online ahead of print. PMID 41324566